CLINICAL TRIAL: NCT04009707
Title: Comparison of 2 Tests for Screening for Cognitive Disorders (MoCA / BEARNI)
Brief Title: Comparison of 2 Tests to Diagnose Cognitive Dysfunctions in Alcohol Disease
Acronym: MoCA/BEARNI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2017/PP-02
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2019-07

CONDITIONS: Alcohol Use Disorder
Keywords: MoCA; BEARNI
MeSH Terms: conditions — Alcoholism | interventions — Mental Status and Dementia Tests; Ethanol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with alcool use desorders: Patient cared for in the addictology department of the University Hospital of Nîmes
  Interventions: Other: MoCA (Montreal Cognitive Assessment) test; Other: BEARNI (Brief Evaluation of Alcohol Related Neuropsychological Impairment) Test

INTERVENTIONS:
Other: MoCA (Montreal Cognitive Assessment) test — the MoCA questionnaire is used to assess cognitive disorders
Other: BEARNI (Brief Evaluation of Alcohol Related Neuropsychological Impairment) Test — This questionnaire is used to assess cognitive disorders

SUMMARY:
The objective of this study is therefore to compare the results obtained with these two screening tests, using as gold standard the results obtained by the battery of neuropsychological reference tests.

DETAILED DESCRIPTION:
Recently, a new screening test for cognitive disorders was specifically developed for patients with UAS: BEARNI (Brief Evaluation of Alcohol-Related Neuropsychological Impairments). Since the BEARNI is presented as the reference test, the investigators have systematically proposed it to hospitalized patients, in combination with the usual check-up. In practice, at admission, patients were therefore given two screening tests, the MoCA and the BEARNI. In the event of an anomaly in at least one of these tests, a battery of confirmatory neuropsychological tests was performed.

ELIGIBILITY:
Inclusion Criteria:

* patients with alcoo use desorder
* Patient cared for in the addictology department of the University Hospital of Nîmes

Exclusion Criteria:

* refusal to use the data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with alcoo use desorder
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
sensitivity | Day 1 (only 1 time)
  comparison of the sensitivity of the 2 tests against the gold standard
specificity | Day 1 (only 1 time)
  comparison of the specificity of the 2 tests against the gold standard

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nîmes, Nîmes, France

REFERENCES:
- [Result] Pelletier S, Alarcon R, Ewert V, Forest M, Nalpas B, Perney P. Comparison of the MoCA and BEARNI tests for detection of cognitive impairment in in-patients with alcohol use disorders. Drug Alcohol Depend. 2018 Jun 1;187:249-253. doi: 10.1016/j.drugalcdep.2018.02.026. Epub 2018 Apr 10. PMID 29684893